CLINICAL TRIAL: NCT01228188
Title: Surgical Inverted ILM Repositioning as Autologous Dressing for Idiopathic Full Thickness Macular Holes Treatment
Brief Title: Inverted ILM Repositioning as Treatment for Full Thickness Macular Holes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Department of Ophthalmology, Military Insitute of Medicine Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BW1127/10
Record Dates: First submitted 2010-10-22; First posted 2010-10-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-09

CONDITIONS: Macular Holes
Keywords: FTMH; PPV; inverted ILM repositioning
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Idiopathic Full Thickness Macular Hole (Experimental): Eyes which do not undergo early vitrectomy at the time of enrollment. Surgical intervention would be performed when full-thickness macular hole occurs with a minimum diameter exceeding 400 um.
  Interventions: Procedure: Inverted ILM Repositioning

INTERVENTIONS:
Procedure: Inverted ILM Repositioning — Three port pars plana vitrectomy is performed by one surgeon (JR). Induction of PVD is initiated by active suction with the vitrectomy probe over the ONH and continued peripherally. First a 0.6-1.0mm piece of ILM surrounding the macular hole is removed. Then significant margin of ILM in macular hole circumference is released while staying connected at the base to the macularrhexis border. Excess of ILM is trimmed. Perfluorocarbon is administrated, stabilizing ILM flap and facilitating the flap repositioning. Trypan Blue is used to stain the ILM. ILM flap is pressed down over the macular hole. The procedure is ended by SF6 gas tamponade. Even in absence of cataract formation, a combined procedure is performed because of exact peripheral vitreous shaving and prevention of cataract formation.
  Other Names: inverted ILM; ILM flap

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of surgical treatment of FTMH using an inverted ILM repositioning to improve anatomical and functional outcomes in patients with a macular hole.

DETAILED DESCRIPTION:
At present, the anatomical closure rate of macular hole is around 90% using pars plana vitrectomy with ILM peeling. Improvement of visual acuity is around 80% including stage II to IV. With macular hole greater than 400 μm there is higher risk of surgical failure and visual acuity is usually less than 0.2. Large macular holes are more likely to have flat-open type closure, which is anatomical success but has limited improvement in visual acuity. Inverted ILM repositioning will form a scaffold for glial cells, which allows their migration and proliferation. This process will close the macular hole and secure it from re-opening, and will reduce the risk of flat-open type of closure.

The aim of this study is to estimate the efficiency and safety of inverted ILM repositioning in the treatment of macular hole with a minimum diameter exceeding 400 μm and compare results with the currently used methods of surgical large macular holes treatment.

ELIGIBILITY:
Inclusion Criteria:

* full-thickness macular hole with a minimum diameter exceeding 400 μm
* BCVA of 0,3 or worse in log MAR units (<=70 ETDRS letter) and 1,6 or better in log MAR units (>=5 ETRDS letter)
* 18 years of age
* Informed consent

Exclusion Criteria:

* eyes with previous vitreous surgery
* cystoid macular edema from any cause
* post traumatic macular hole
* macular hole associated with retinal detachment
* any other ocular reason which causes the lack of improvement after macular hole surgery (e.g pigmentary abnormalities, age-related macular degeneration, corneal scarring)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA), postoperative macular hole closure type | up to 1 week before surgery
  BCVA for ETDRS chart (converted to logMAR) and postoperative macular hole closure type assessed by OCT: elevated-open, flat-open and flat-closed.
Best-corrected visual acuity (BCVA), postoperative macular hole closure type | 2 weeks postoperatively ( plus or minus 1 week)
  BCVA for ETDRS chart (converted to logMAR) and postoperative macular hole closure type assessed by OCT: elevated-open, flat-open and flat-closed.
Best-corrected visual acuity (BCVA), postoperative macular hole closure type | 4 weeks postoperatively ( plus or minus 1 week)
  BCVA for ETDRS chart (converted to logMAR) and postoperative macular hole closure type assessed by OCT: elevated-open, flat-open and flat-closed.
Best-corrected visual acuity (BCVA), postoperative macular hole closure type | 6 weeks postoperatively ( plus or minus 1 week)
  BCVA for ETDRS chart (converted to logMAR) and postoperative macular hole closure type assessed by OCT: elevated-open, flat-open and flat-closed.
Best-corrected visual acuity (BCVA), postoperative macular hole closure type | 12 weeks postoperatively ( plus or minus 1 week)
  BCVA for ETDRS chart (converted to logMAR) and postoperative macular hole closure type assessed by OCT: elevated-open, flat-open and flat-closed.
Best-corrected visual acuity (BCVA), postoperative macular hole closure type | 24 weeks postoperatively ( plus or minus 1 week)
  BCVA for ETDRS chart (converted to logMAR) and postoperative macular hole closure type assessed by OCT: elevated-open, flat-open and flat-closed.
Best-corrected visual acuity (BCVA), postoperative macular hole closure type | 48 weeks postoperatively ( plus or minus 1 week)
  BCVA for ETDRS chart (converted to logMAR) and postoperative macular hole closure type assessed by OCT: elevated-open, flat-open and flat-closed.

SECONDARY OUTCOMES:
Central Macular Thickness (CMT), Central Macular Volume | up to 1 week before surgery
  Central Macular Thickness (CMT)and Central Macular Volume are assessed 1 mm and 6 mm diameter topography (OCT-SLO).
Central Macular Thickness (CMT), Central Macular Volume | 2 weeks postoperatively (plus and minus 1 week)
  Central Macular Thickness (CMT)and Central Macular Volume are assessed 1 mm and 6 mm diameter topography (OCT-SLO).
Central Macular Thickness (CMT), Central Macular Volume | 4 weeks postoperatively (plus and minus 1 week)
  Central Macular Thickness (CMT)and Central Macular Volume are assessed 1 mm and 6 mm diameter topography (OCT-SLO).
Central Macular Thickness (CMT), Central Macular Volume | 6 weeks postoperatively (plus and minus 1 week)
  Central Macular Thickness (CMT)and Central Macular Volume are assessed 1 mm and 6 mm diameter topography (OCT-SLO).
Central Macular Thickness (CMT), Central Macular Volume | 12 weeks postoperatively (plus and minus 1 week)
  Central Macular Thickness (CMT)and Central Macular Volume are assessed 1 mm and 6 mm diameter topography (OCT-SLO).
Central Macular Thickness (CMT), Central Macular Volume | 24 weeks postoperatively (plus and minus 1 week)
  Central Macular Thickness (CMT)and Central Macular Volume are assessed 1 mm and 6 mm diameter topography (OCT-SLO).
Central Macular Thickness (CMT), Central Macular Volume | 48 weeks postoperatively (plus and minus 1 week)
  Central Macular Thickness (CMT)and Central Macular Volume are assessed 1 mm and 6 mm diameter topography (OCT-SLO).

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Robaszkiewicz, dr med., Principal Investigator — Department of Ophthalmology Military Institute of Medicine
Locations (1):
- Military Institute of Medcine, Warsaw, Ul. Szaserów 128, Poland